CLINICAL TRIAL: NCT04523337
Title: A Randomized Controlled Trial of MISSION-CJ for Justice-Involved Homeless Veterans With Co-Occurring Substance Use and Mental Health Disorders
Brief Title: MISSION-CJ for Justice-Involved Homeless Veterans
Acronym: MISSION-CJ
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 18-040
Record Dates: First submitted 2020-07-28; First posted 2020-08-21 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Substance Use Disorder; Mental Health Disorder; Homelessness
Keywords: Veterans; Co-Occurring Disorder; Homeless Persons; crime; substance-related disorders; mental disorders
MeSH Terms: conditions — Substance-Related Disorders; Mental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Research assistants conducting the 6- and 15-month outcome assessments are blinded to the condition assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MISSION-CJ (Experimental): Maintaining Independence and Sobriety through Systems Integration Outreach and Networking- Criminal Justice version (MISSION-CJ) programming targets co-occurring substance use and mental health disorders and other related health outcomes faced by justice-involved homeless Veterans through assertive outreach, psychoeducation, and linkages to community-based services.
  Interventions: Behavioral: Maintaining Maintaining Independence and Sobriety through Systems Integration Outreach and Networking- Criminal Justice
- Enhanced Usual Care (Experimental): Usual care provided by the mental health residential rehabilitation treatment programs, with patients in both groups are enrolled in, in addition to peer support and community outreach case management. Patients receive 2 Peer Support Curriculum sessions per week (24 sessions total). Patients will receive unstructured community outreach and linkage support while enrolled in the mental health residential rehabilitation program. After discharge, patients will continue to receive 1 hour of weekly linkage support per week.
  Interventions: Behavioral: Maintaining Maintaining Independence and Sobriety through Systems Integration Outreach and Networking Peer Support

INTERVENTIONS:
Behavioral: Maintaining Maintaining Independence and Sobriety through Systems Integration Outreach and Networking- Criminal Justice — Maintaining Independence and Sobriety through Systems Integration Outreach and Networking- Criminal Justice version (MISSION-CJ) programming targets co-occurring substance use and mental health disorders and other related health outcomes faced by justice-involved homeless Veterans through assertive outreach, psychoeducation, and linkages to community-based services. Patients will receive 2 hours of MISSION-CJ services per week during and after their stay in the mental health residential rehabilitation program (total of 6-months). Services are delivered using a Critical Time Intervention stepdown approach.
  Other Names: MISSION-CJ
  Arms: MISSION-CJ
Behavioral: Maintaining Maintaining Independence and Sobriety through Systems Integration Outreach and Networking Peer Support — The MISSION Peer Support Curriculum is rolling entry, and includes 24, one-hour exercises focused on co-occurring substance use and mental health disorders, recovery, and community integration.
  Other Names: MISSION Peer Support
  Arms: Enhanced Usual Care

SUMMARY:
The purpose of this study is to determine whether Maintaining Independence and Sobriety through Systems Integration, Outreach and Networking - Criminal Justice version (MISSION-CJ) is effective for reducing criminal recidivism and improving other health-related outcomes (substance use, mental health, housing, employment, community integration) among justice-involved, homeless Veterans with a co-occurring substance use and mental health disorder.

DETAILED DESCRIPTION:
VHA Mental Health Residential Rehabilitation Treatment Programs (MH RRTPs) serve Veterans with an estimated 50% having criminal justice involvement annually. Justice-involved Veterans (JIVs) receive assistance with their addiction and behavioral health needs, but MH RRTP programs do not directly address their antisocial behaviors and cognitions. Furthermore, MH RRTP discharge is a vulnerable transition and no national transitional approach facilitates Veteran's engagement in prosocial community behaviors that sustain MH RRTP gains, ultimately reducing revolving door service use.

Maintaining Independence and Sobriety through Systems Integration, Outreach, and Networking-Criminal Justice version (MISSION-CJ) is a new case manager and peer delivered team-based treatment for JIVs with a co-occurring substance use and mental health disorder (COD). While MISSION-CJ derives in part from an evidence-based treatment for homeless individuals (MISSION), it includes a new conceptual framework and numerous new and differentiating features for a CJ population including: (1) a treatment planning tool focused on criminogenic needs that monitors progress and tunes service delivery elements; (2) a prosocial treatment curriculum; and (3) tools/resources to address JIVs' legal issues. With MISSION-CJ, this study attempts to change the practice paradigm and transform care for JIVs by moving beyond the current model of linking Veterans to VA care and tracking behavioral health outcomes, to a hybrid treatment/linkage approach that addresses criminogenic needs, supports engagement in VA and non-VA care, and targets recidivism as an outcome-the gold standard for CJ research.

Using a Hybrid Type 1 design, this project will test the effectiveness of MISSION-CJ in a three-site RCT (Bedford, Palo Alto, and Little Rock VAs) with JIVs with a COD, admitted to an MH RRTP, and previously arrested and charged and/or released from incarceration in the past 5-years.

ELIGIBILITY:
Inclusion Criteria:

* (a) are entering a Mental Health Residential Rehabilitation Treatment Program (MH RRTP)
* (b) were arrested and charged and/or released from incarceration in the past 5 years
* (c) have a co-occurring substance use and mental health disorder (COD)

Exclusion Criteria:

* The only exclusion criterion is being too cognitively impaired to understand the informed-consent process and other study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Criminal recidivism | through study completion, on average 15-months
  Number of arrests based on records from the California and Massachusetts Department of Corrections records; and arrest and incarceration records from the National Crime Information Center.
Criminal recidivism | through study completion, on average 15-months
  Number of charges based on records from the California and Massachusetts Department of Corrections records; and arrest and incarceration records from the National Crime Information Center.
Criminal Recidivism | through study completion, on average 15-months
  Number of nights in jail or prison based on records from the California and Massachusetts Department of Corrections records; and arrest and incarceration records from the National Crime Information Center.

SECONDARY OUTCOMES:
Change in Substance use (Alcohol Use Timeline Follow-back -TLFB) | Baseline, 6-months, 15-months
  Quantity of patients' self-reported alcohol use in the past 90 days. Frequency and quantity will be combined to measure alcohol use severity.
Change in Substance use (Alcohol Use Timeline Follow-back -TLFB) | Baseline, 6-months, 15-months
  Frequency of patients' self-reported alcohol use in the past 90 days. Frequency and quantity will be combined to measure alcohol use severity.
Change in Substance Use (Illicit Drug Use Timeline Follow back - TLFB) | Baseline, 6-months, 15-months
  Quantity of patients' self-reported illicit drug use in the past 90 days. Frequency and quantity will be combined to measure drug use severity.
Change in Substance Use (Illicit Drug Use Timeline Follow back - TLFB) | Baseline, 6-months, 15-months
  Frequency of patients' self-reported illicit drug use in the past 90 days. Frequency and quantity will be combined to measure drug use severity.
Change in Trauma Symptoms (PTSD Checklist for DSM-5 - PCL-5) | Baseline, 6-months, 15-months
  Changes in the severity of patients' PTSD symptoms. A total severity score is computed by summing all the items. Scores range from 0-80 with higher scores indicating higher severity.
Change in Depression (Patient Health Questionnaire-9 - PHQ-9) | Baseline, 6-months, 15-months
  Changes in the degree of depression severity self-reported by patients. Total scores range from 0-27 with higher scores indicating more severe depression.
Change in Mental Health Symptoms (Behavior and Symptom Identification Scale-24 - BASIS-24) | Baseline, 6-months, 15-months
  Changes in the severity of patients' self-reported psychiatric symptoms across 6 subscales (e.g. Depression and Functioning, Interpersonal Relationships, Self-Harm, Psychosis, Substance Abuse, and Emotional Lability) during the past week. Patients score items on a scale of 0-4, and each subscale and mean total score range from 0-4, with higher scores indicating higher levels of severity of symptoms.
Change in Recidivism risk (Level of Service Inventory-Revised) | Baseline, 6-months, 15-months
  Changes in the severity of patients' self-reported legal problems. Self-reported arrests, charges, and months incarcerated since the baseline assessment. Total LSI-R scores will be used. Scores range from 0-54 with higher scores indicating greater risk.
Change in Medication Adherence Rating Scale (MARS) | Baseline, 6-months, 15-months
  Patients' self-reported compliance with medication. Questions are dichotomous yes/no.
Change in Housing Status (Residential Timeline Follow back) | Baseline, 6-months, 15-months
  Quantity of patients' self-reported days homeless in the past 90 days.
Change in Housing Status (Residential Timeline Follow back) | Baseline, 6-months, 15-months
  Frequency of patients' self-reported days homeless in the past 90 days.
Change in Employment (Maudsley Addiction Profile) | Baseline, 6-months, 15-months
  Quantity of days worked, days absent, and days unemployed in the past 30 days, as self-reported by patients since the baseline assessment.
Change in Employment (Maudsley Addiction Profile) | Baseline, 6-months, 15-months
  Frequency of days worked, days absent, and days unemployed in the past 30 days, as self-reported by patients since the baseline assessment.
Treatment Engagement (MISSION Treatment Services Tracking Sheet | Up to 12 months
  Number of services for both VA and non-VA services received (pre- and post-MH RRTP). This includes all possible services offered within MISSION-CJ and EUC (MISSION Peer Support) as well as community linkages. Regarding linkages, the measure quantifies the number of referrals, referral type, and client engagement. Examine change in number of services received during 12 months, collected on a weekly basis.
Treatment Engagement (MISSION Treatment Services Tracking Sheet) | Up to 12 months
  Types of services for both VA and non-VA services received (pre- and post-MH RRTP). This includes all possible services offered within MISSION-CJ and Enhanced Usual Care (MISSION Peer Support) as well as community linkages. Examine change in types of services received during 12 months, collected on a weekly basis.
Change in Treatment Engagement (Alcoholics Anonymous Involvement Scale - AAI) | Baseline, 6-months, 15-months
  Change in patients' self-reported involvement in 12-step groups for substance use. Items are dichotomous yes/no, with yes responses indicating more involvement in 12-step groups. Composite scores range from 0-9 with 9 indicating more involvement in 12-step groups. Patients are also asked to indicate which of the 12-steps they have worked.
Change in Treatment Engagement (Alcoholics Anonymous Involvement Scale - AAI) | Baseline, 6-months, 15-months
  Change in patients' self-reported attendance in 12-step groups for substance use over lifetime, and since the previous assessment. Patients report an estimated number of meetings they've attended in the last year, and in their lifetime.
Treatment Engagement (Healthcare Continuing Care Utilization) | 12-month period prior to, and ending 15 months after, study enrollment
  Data on SUD/MH continuing care utilization since the prior assessment will be defined as the number of sessions in each setting that the clients attend throughout the follow-up period. Both will be obtained from: (a) CDW, for VA care and (b) service tracking sheets for VA and non-VA health care utilization. For VA care, the electronic medical record data will be obtained from the CDW. CDW data includes both outpatient encounter records (including the type of outpatient care - e.g., from outreach programs, office-based clinical services) and information on inpatient and residential care services used.
Treatment Engagement (MH RRTP Completion) | 12-month period prior to, and ending 15 months after, study enrollment
  Healthcare utilization includes both VA and non-VA healthcare services and we will construct several measures. MH RRTP completion will be defined as a regular discharge from the program and determined from the VA's Corporate Data Warehouse (CDW).
Change in Community Integration Measure (CIM) | Baseline, 6-months, 15-months
  Patient's self-report perspective of their integration into their home and community are scored on a 5-point scale. A single summary score (range 10-50) is computed by summing each item, with lower scores indicating
Change in Antisocial Attitudes (Measures of Criminal Attitudes and Associates - MCAA) | Baseline, 6-months, 15-months
  Changes in patients' self-report of antisocial attitudes on 4 scales: violence, entitlement, antisocial intent, and associates. Responses to MCAA Part B are dichotomous agree/disagree.
Change in Affiliations with Antisocial Peers (Measures of Criminal Attitudes and Associates: MCAA) | Baseline, 6-months, 15-months
  Changes in patients' self-report of criminal associations. Part A of the MCAA is intended to quantify criminal associations. In Part A, respondents are asked to recall the four adults in the community with whom they spend the most free time. For each adult, they then indicate how much of their free time is spent in their associate's company. The respondent then answers four questions regarding the degree of criminal involvement of their associates: (a) Has this person ever committed a crime; (b) Does this person have a criminal record; (c) Has this person ever been to jail? and (d) Has this person tried to involve you in a crime? From this information, a measure of criminal associates can be calculated. The Number of Criminal Friends is calculated by totaling the number of friends for which the respondent answers yes to any of the questions of criminal involvement.

CONTACTS AND LOCATIONS:
Overall Officials: David A. Smelson, PsyD, Principal Investigator — VA Bedford HealthCare System, Bedford, MA; Daniel M. Blonigen, PhD MA, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (3):
- United States (3):
  - Central Arkansas VHS John L. McClellan Memorial Veterans Hospital, Little Rock, AR, Little Rock, Arkansas
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - VA Bedford HealthCare System, Bedford, MA, Bedford, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shaffer PM, Andre M, Smelson D, Cucciare MA, Bruzios KE, Blonigen DM. Criminogenic risk and suicidality among justice-involved homeless veterans with comorbid mental health and substance use disorders. BMC Public Health. 2026 Feb 4. doi: 10.1186/s12889-026-26250-6. Online ahead of print. PMID 41639846
- [Derived] Bruzios K, Shaffer PM, Blonigen DM, Cucciare MA, Andre M, Byrne T, Smith J, Smelson D. Intervention for Justice-Involved Homeless Veterans With Co-Occurring Substance Use and Mental Health Disorders: Protocol for a Randomized Controlled Hybrid Effectiveness-Implementation Trial. JMIR Res Protoc. 2025 Jul 18;14:e70750. doi: 10.2196/70750. PMID 40680272